CLINICAL TRIAL: NCT06025630
Title: Targeting Endoplasmic Reticulum Stress in Human Hypertension
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Principal Investigator, Steven A. Romero, Associate Professor, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ERX:2023-063
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
Keywords: high blood pressure; tauroursodeoxycholic acid (TUDCA); endoplasmic reticulum
MeSH Terms: conditions — Hypertension | interventions — ursodoxicoltaurine

STUDY DESIGN:
Intervention Model Description: This study uses a single-blind, placebo-controlled model.
Who Masked: Participant
Masking Description: Participants will be blinded to which condition they are randomly assigned (placebo vs TUDCA ingestion)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoplasmic Reticulum Stress Inhibition (Experimental)
  Interventions: Drug: TUDCA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TUDCA — Endoplasmic reticulum stress will be inhibited by chronic (8 weeks) oral ingestion of the dietary supplement tauroursodeoxycholic acid (TUDCA; 1,750 mg/day)
  Arms: Endoplasmic Reticulum Stress Inhibition
Drug: Placebo — Placebo pills containing microcrystalline cellulose will be ingested over the course of the 8 week intervention.
  Arms: Placebo

SUMMARY:
There is strong evidence suggesting that endoplasmic reticulum stress contributes to neurogenic and vascular hypertension in various animal models, however this has never been explored in humans. Therefore, this project will fill this gap by performing a single-blind, placebo-controlled trial in humans with hypertension.

DETAILED DESCRIPTION:
The endoplasmic reticulum is a multipurpose organelle found in most human cells, including those in the brain and the endothelium of blood vessels. One of the primary functions of the endoplasmic reticulum is the posttranslational folding of new proteins and the reprocessing of misfolded or damaged proteins. Physiological and pathophysiological conditions can lead to the accumulation of unfolded/misfolded proteins, thus triggering the unfolded protein response which is a quality control system that maintains endoplasmic reticulum homeostasis. However, with prolonged or severe exposure to endoplasmic reticulum stress inducers, the unfolded protein response can augment the formation of reactive oxygen species, inflammatory mediators, and transcription factors that trigger sympathetic overactivity and induce endothelial dysfunction. There is strong evidence suggesting that endoplasmic reticulum stress contributes to neurogenic and vascular hypertension in various animal models, however this has never been explored in humans. This proposal builds on prior work in which the investigators pharmacologically augmented circulating concentrations of the potent endoplasmic reticulum stress inhibitor, tauroursodeoxycholic acid (TUDCA) and the development of an assay/test to quantify endoplasmic reticulum stress in cutaneous biopsy samples.

This study will accomplish the following Specific Aims:

1. Examine if endoplasmic reticulum stress inhibition, via chronic ingestion of tauroursodeoxycholic acid, will attenuate 24h blood pressure in humans with elevated (120-129/<80 mmHg) or stage 1 (130-140/80-90 mmHg) hypertension.
2. Examine the extent to which endoplasmic reticulum stress inhibition alters neurovascular control in the participants of Aim 1. Independent of the contribution to blood pressure regulation, neurovascular function is considered a key risk factor for cardiovascular morbidity and mortality. As such, the outcome of Aim 2, while providing mechanistic insight into the blood pressure lowering effect of endoplasmic reticulum stress inhibition, should be considered independent of the outcomes of Aim 1.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age
2. No tobacco/nicotine use within preceding 6 months (e.g., cigarettes, chewing tobacco, nicotine gum or patches)
3. Systolic blood pressure <140 mmHg; diastolic blood pressure <90 mmHg (obtained at the Screening and Familiarization Visit)
4. Normal 12-lead ECG (obtained at the Screening and Familiarization Visit and reviewed by a board-certified physician)
5. Normal clinical results from a medical exam reviewed by a board-certified physician (e.g., General Health Questionnaire obtained at the Screening and Familiarization Visit)
6. Body mass index (BMI) <35 unless athletic/muscular build; calculation = body weight (kg)/height (m2);
7. Females only: documentation of a negative pregnancy test prior to the familiarization and experimental sessions unless post-menopausal

Exclusion Criteria:

1. Not meeting the defined age criteria
2. Body mass index (BMI) >35 unless athletic/muscular build; calculation = body weight (kg)/height (m2)
3. Any tobacco/nicotine use within the last 6 months (e.g., cigarettes, chewing tobacco, nicotine gum or patches)
4. Positive pregnancy test
5. Females with an erratic/irregular menstrual cycle
6. Females who are breastfeeding
7. Women who are prescribed a continually releasing hormonal contraceptive (e.g. NuvaRingTM or other hormone releasing vaginal rings, Depo Provera shot, or birth control implants such as Nexplanon)
8. Subjects who weigh less than 80 lbs.
9. Use of prescription drugs, non-prescription drugs, dietary supplements or herbal medicines known to alter vascular function unless cleared prior to the study
10. Use of beta blockers
11. Daily use of bronchodilators
12. Use of anti-coagulant therapy
13. Implanted medical devices (e.g. cardiac pacemaker)
14. Current or past history of hyperthyroidism, or other thyroid hormone-related disease
15. Current use of hormone replacement therapy (e.g., estrogen, testosterone)
16. HbA1c >5.6
17. Resting systolic blood pressure of <100 mmHg; >140mmHg or diastolic blood pressure >90mmHg
18. Abnormal 12-lead ECG or uncontrolled heart rhythm issues causing symptoms, or an unstable blood pressure
19. History of cerebrovascular abnormalities (e.g., prior stroke, transient ischemic attacks, epilepsy)
20. Known history of atherosclerosis of the carotid arteries (i.e., plaque formation)
21. History of concussion and or other loss of consciousness within the preceding 30 days
22. Autonomic dysfunction (e.g., Shy-Drager Syndrome, Bradbury-Eggleston syndrome, sinus arrhythmia, idiopathic orthostatic hypotension, fainting disorder)
23. Respiratory illnesses (e.g., chronic asthma (including exercise-induced asthma), Chronic Obstructive Pulmonary Disease, Reactive Airway Disease)
24. Any prior history of anaphylaxis, not just prior reactions to the materials used in this study
25. Severe phobia of needles
26. Latex allergy aa) Known allergies or sensitivities to substances used in the study (e.g., Lidocaine HCL, sodium nitroprusside, acetylcholine, phentolamine, L-NAME, TUDCA, or related drugs) bb) Donated blood within the last 60 days cc) History or family history of abnormal blood clotting, clots in deep veins in the legs or pelvis, or blood clots to the lungs dd) History of alcohol or drug abuse which inhibits the subject's ability to complete this study ee) Individuals who have had mastectomies ff) History of methemoglobinemia gg) Current diagnosis of anemia hh) Current Fever (oral temp >99.5 °F/ 37.5 °C) ii) Current use of PDE3 inhibitors (e.g., Viagra) or soluble guanylate cyclase (sGC) stimulators (e.g., riociguat), or unwillingness to withhold medication for 2 weeks prior to laboratory testing jj) Current diagnosis of cancer kk) Cardiac surgery or cardiac events (e.g., coronary artery bypass graft surgery, myocardial infarction, heart failure) ll) Diagnosis of neurological disease or cognitive dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
24 hour Blood Pressure | Within 1-2 weeks before and after intervention or placebo
  Systolic and diastolic blood pressure will be measured twice per hour during the day and once per hour at night using a portable cuff.

SECONDARY OUTCOMES:
Neurovascular Function | Within 1-2 weeks before and after intervention or placebo
  The microdialysis technique will be used to examine neurovascular function. To do this, blood flow will be measured in response to the local infusion of pharmacological agents that alter blood flow.
Cardiac output | Within 1-2 weeks before and after intervention or placebo
  The amount of blood pumped from the heart each minute (i.e., cardiac output) be measured via inert gas (nitrous oxide) rebreathing
Arterial Pulse Wave Velocity | Within 1-2 weeks before and after intervention or placebo
  Resting arterial compliance/stiffness will be assessed by measuring Doppler derived pulse wave velocity.
Endoplasmic Reticulum Stress | Within 1-2 weeks before and after intervention or placebo
  Endoplasmic reticulum stress will be quantified by measuring the mRNA expression of spliced X-box binding protein 1 in a cutaneous biopsy sample obtained before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No